CLINICAL TRIAL: NCT04858308
Title: Phase 3 Trial to Evaluate the Efficacy and Safety of YYC506.
Acronym: Atorf-YOOrct
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yooyoung Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YYPCT_YYC506_301
Record Dates: First submitted 2021-04-20; First posted 2021-04-26 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Dyslipidemias
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Intervention Model Description: A multicenter, Double-blind, Randomized, Active-controlled, Double dummy, Parelle-group comparative.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Active Comparator): Take both YYC506 and Placebo(Control)
  Interventions: Drug: YYC506; Drug: Control Placebo
- Control Group (Active Comparator): Take both Contral and Placebo(YYC506)
  Interventions: Drug: Control; Drug: YYC506 Placebo

INTERVENTIONS:
Drug: YYC506 — YYC506
  Arms: Test Group
Drug: Control — Active control
  Arms: Control Group
Drug: YYC506 Placebo — Placebo
  Arms: Control Group
Drug: Control Placebo — Placebo
  Arms: Test Group

SUMMARY:
Phase 3 study to evaluate the effiacay and safety of YYC506

DETAILED DESCRIPTION:
Phase 3 study to evaluate the effiacay and safety of YYC506 in patients with complex dyslipidemia where LDL-C is properly controlled but TG and HDL-C levels are not regulated by Atorvastatin alone.

ELIGIBILITY:
Inclusion Criteria:

* A man or woman over 19 years old.
* LDL-C properly controlled, TG, HDL-C is not properly controlled
* Sign on ICF prior to study participation

Exclusion Criteria:

* History of Fibromyalgia, Myopathy etc (CK ≥ 2XULN)
* Uncontrolled hypo-thyroidism (TSH≥1.5XULN)
* Severe renal impairemnet (Creainine clearance < 30mL/min) etc.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 554 (Estimated)
Dates: Start 2021-01-29 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Percent change (%) of non-HDL-C from baseline | from baseline at 12 weeks
  non HDL-C = TC - HDL-C

SECONDARY OUTCOMES:
Percent change (%) of non-HDL-C | from baseline at 4, 8, 14 weeks.
  non HDL-C = TC - HDL-C
Percent change (%) of lipid parameters | from baseline at 4, 8, 12, 24 weeks
  TC, HDL-C, LDL-C, TG
Percent change (%) of diabetes parameters | from baseline at 4, 8, 12, 24 weeks
  FBS, HbA1c, Insulin

CONTACTS AND LOCATIONS:
Overall Officials: Hyo-soo Kim, Ph.D, Study Chair — Seoul National University Hospital; Hyo-soo Kim, Ph.D, Principal Investigator — Seoul National University Hospital; Soo Lim, Ph.D, Principal Investigator — Seoul National University Bundang Hospital
Locations (3):
- South Korea (3):
  - Chonbuk National University Hospital, Cheonju
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National UniversityHospital, Seoul

IPD SHARING:
Plan to Share IPD: No